CLINICAL TRIAL: NCT02341768
Title: Clinical and Device Functional Assessment of Real World ICD Patients
Acronym: CARAT
Status: Completed | Type: Observational
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Other Study IDs: RTSY03
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Arrythmia; Implantable Cardioverter Defibrillator
Keywords: clinical and device functional information; "real world" ICD patient population
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ICD — ICD single, dual or triple chamber, upgrade, replacement or primo implant

SUMMARY:
The primary requirement of the implantable cardioverter defibrillator (ICD) is to preserve life by terminating life-threatening arrhythmias (VT/VF). The treatment options vary in terms of techniques and medical devices, based on the patient's condition.

It is extremely important in the clinical practice to identify which patients' subgroup benefits the most from the ICD therapy, which comorbidity has a major impact on the patients' prognosis, or which pre-intra-post procedural behaviors provoke less complications, and affect the patient's outcome (including prolonged or unwanted hospitalizations).

DETAILED DESCRIPTION:
For these reasons, it is very important to observe the clinical practice on a large variety of centers and countries, with the objective to collect long term safety and performance data in patients undergoing ICD/CRT-D device implantation (first implant, replacement or upgrade).

The safety and performance of the ICDs can be evaluated through the collection of multiple parameters such as, but not limited to:

* Clinical parameters, like patient demographics and history, procedural and hospital discharge data, as well as the short and long term serious adverse events (death and hospitalization)
* Device parameters, such as delivered shocks, ATP, or other device therapies

Worldwide selected centers will be invited to participate in this prospective study and include their "real-world" patients treated with Sorin Group commercially available ICDs and CRT-Ds devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient Implanted (first implant, replacement, upgrade) with a Sorin Group ICD/CRT-D device, according to current available guidelines and IFU
* Signed and dated informed consent (in accordance to local regulation)

Exclusion Criteria:

* Already included in another clinical study that could confound the results of this study
* Not available for routine follow-up visits
* Minor age
* Drug addiction or abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to include all patients from a global "real world" (standard of care) population at participating centers and will reference the indication and the contra-indications specified in the guidelines and IFUs.
Sampling Method: Non-Probability Sample
Enrollment: 2056 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Evaluate clinical and device functional information from "real world" ICD patient population following standard of care at participating centers w/in the different participating countries (Incidence of all death, device,cardiac related hospitalization) | 2 years
  Incidence of all death, device and/or cardiac related hospitalization at 24 months post implant

SECONDARY OUTCOMES:
Serious procedural complications or other SAE at implantation or hospital discharge. The data analyzed are those collected from the day of implantation to the day of hospital discharge, with an expected average of 1 week. | at implantation or hospital discharge
  as reported by the sites on the AE eCRF
The incidence of all death, device and/or cardiac related hospitalization at 12 months post implant (evaluated with a survival curve) | at 12 months
  as reported by the sites with AE
The predictors of mortality and cardiac related hospitalization at 12 and 24 months | at 12 and 24 months
  as reported by the sites with AE and medical history information
The predictors of appropriate or inappropriate therapies (ATP and shocks) at 12 and 24 months, as verified by a dedicated committee | at 12 and 24 months
  based on therapies delivered recorder on device file, and verified by a dedicated committee
The evolution of the indication for implant according to guideline (based on the patient's medical history and reason for implant as reported by the investigators) | at implant
  based on the patient's medical history and reason for implant as reported by the investigators

CONTACTS AND LOCATIONS:
Overall Officials: Javier Moreno, Dr, Principal Investigator — Hospital Ramón y Cajal Ctra. de Colmenar Viejo km 9.100, 28034 Madrid, Spain
Locations (102):
- Austria (4):
  - LKH Feldkirch, Feldkirchen bei Mattighofen
  - LKH Innsbruck, Innsbruck
  - Kepler Universitatsklinikum GmbH, Linz
  - LKH St. Polten, Pölten
- Canada (6):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Royal Alexandra Hospital, Edmonton
  - HDM (CHUM) Montreal, Montreal
  - HSCM Montreal, Montreal
  - IUCPQ Quebec, Québec
  - Sherbrooke, Québec
- Czechia (3):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice U svaté Anny v Brno, Brno
  - Fakultni Nemocnice Olomouc, Olomouc
- France (32):
  - CHU Angers, Angers
  - CH Annecy Genevois, Annecy
  - Clinique Rhône Durance, Avignon
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - H.I.A Percy, Clamart
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CH de Marne la Vallée, Jossigny
  - Hôpital Louis Pasteur, Le Coudray
  - CHRU de Lille, Lille
  - CH St Joseph St Luc, Lyon
  - Hôpital la Timone, Marseille
  - Hôpital Nord Marseille, Marseille
  - Hôpital Jacques Cartier, Massy
  - CHU A de Villeneuve, Montpellier
  - Clinique du Millénaire, Montpellier
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU de Nimes, Nîmes
  - HEGP, Paris
  - La Pitié Salpétrière, Paris
  - CHU François Mitterand, Pau
  - CH Perpignan, Perpignan
  - CHU de Poitiers, Poitiers
  - CHRU de Pontchaillou, Rennes
  - CHRU de Rouen, Rouen
  - CHU de Valence, Valence
  - CH de Villefranche sur Saone, Villefranche-sur-Saône
- Germany (15):
  - Kardiologische Praxis, Altentreptow
  - HGZ Bad Bevensen, Bad Bevensen
  - Herz- und Diabeteszentrum, Bad Oeynhausen
  - Evangelisches Krankenhaus, Bielefeld
  - Universitatskliniken, Bonn
  - Kardiologie Darmstadt, Darmstadt
  - Universitatskliniken Düsseldorf, Düsseldorf
  - Albertinen-Krankenhaus, Hamburg
  - Cardiologicum Hamburg, Hamburg
  - Universität Kiel, Kiel
  - Universitaetsklinikum Schleswig Holstein, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Kardiologische Praxis, Markkleeberg
  - Dietrich Bonhoeffer Klinikum, Neubrandenburg
  - Universitatsklinikum, Würzburg
- Italy (11):
  - Ospedale Garibaldi Centro, Catania
  - Ospedale Pol SS Annunziata, Chieti
  - Presidio Ospedaliero di Chioggia, Chioggia
  - Ospital San Luca, Lucca
  - Ospedale Civile, Mirano
  - Osp S Giovanni Bosco, Napoli
  - Ospedale Cardarelli, Napoli
  - Ospedale Policlinico Federico II, Napoli
  - Policlinico Casilino, Rome
  - Osp. G. Mazzini, Teramo
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Trieste
- Netherlands (2):
  - Vlietland Ziekenhuis, Schiedam
  - Isala Klinieken, Zwolle
- Portugal (4):
  - Hospital Garcia de Orta, Almada
  - Hospital Professor Doutor Fernando Fonseca, Amadora
  - CHLC Hospital de Santa Marta, Lisbon
  - H. Santa Maria, Lisbon
- Slovakia (3):
  - Susch Hospital, Banská Bystrica
  - Nusch Hospital, Bratislava
  - Vusch Hospital, Košice
- Spain (11):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Llàtzer, Palma de Mallorca
  - Complejo Hospitalario Universitario, Santiago de Compostela
  - H.U La Fe, Valencia
  - CHU de Vigo, Vigo
- Fondazione Cardiocentro Ticino, Lugano, Switzerland
- United Kingdom (10):
  - Barnet General Hospital, Barnet
  - Edgbaston, Birmingham
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Dorget County Hospital, Dorchester
  - Royal Infirmary of Edinburgh, Edinburgh
  - Wye Valley NHS Trust, Hereford
  - Glenfield Hospital, Leicester
  - King's College Hospital, London
  - Northampton General Hospital, Northampton
  - Northern General Hospital, Sheffield